CLINICAL TRIAL: NCT07333833
Title: Development and Validation of an Early Prediction Model for Severe Mycoplasma Pneumoniae Pneumonia in Children
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: V120250926
Record Dates: First submitted 2025-12-22; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2018-01

CONDITIONS: Mycoplasma Pneumoniae Pneumonia
Keywords: severe mycoplasma pneumoniae pneumonia
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Development: A primary cohort of eligible patients from the Beijing Friendship Hospital between 2018-1-1 and 2024-5-31 is used for model derivation.
  Interventions: Other: medical history taking, blood test, pulmonary ultrasound
- Internal cross-validation: A cohort of consecutive patients from the Beijing Friendship Hospital between 2018-1-1 and 2024-5-31 is used for internal cross-validation.
  Interventions: Other: medical history taking, blood test, pulmonary ultrasound
- External validation: A cohort of patients from the Beijing Friendship Hospital between 2024-6-1 and 2025-6-30 is used for internal cross-validation.
  Interventions: Other: medical history taking, blood test, pulmonary ultrasound

INTERVENTIONS:
Other: medical history taking, blood test, pulmonary ultrasound — medical history taking, blood test, pulmonary ultrasound are used for MPP and SMPP diagnosis

SUMMARY:
Pneumonia is a major threat to the health of children. Mycoplasma pneumoniae infection is a core cause of pediatric pneumonia, and the incidence of severe mycoplasma pneumoniae pneumonia (SMPP) has increased in recent years. SMPP leads to a range of extrapulmonary symptoms, including myocardial and liver injury, which may be life-threatening. Therefore, there is an urgent need to establish an early warning model for SMPP to improve the prognosis of pediatric pneumonia. This observational study aims to establish a early prediction model of SMPP. Development cohorts are enrolled from Beijing Friendship Hospital between 2018-1-1 to 2024-5-31, and validation cohorts are enrolled between 2024-6-1 to 2025-6-30.

ELIGIBILITY:
Inclusion Criteria:

* Age between 1 month to 14 years
* diagnosed with Mycoplasma pneumoniae pneumonia
* hospital stay ≥ 72 hours

Exclusion Criteria:

* pulmonary chronicles
* cardiovascular conditions
* inherited metabolic disorders
* immuno-deficiency disorders
* coinfection with pathogens other than Mycoplasma pneumoniae

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children hospitalized at Beijing Friendship Hospital between 2018-01-01 and 2024-06-01, diagnosed with MPP, and with a hospital stay > 3 days (aged 1 month to 14 years) were enrolled. According to disease severity, they were divided into the mild MPP (MPP group) and severe MPP (SMPP group).
Sampling Method: Non-Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | through the hospitalization, an average of 7 days
  The AUC of prediction model for SMPP

SECONDARY OUTCOMES:
Sensitivity | through the hospitalization, an average of 7 days
  The sensitivity of prediction model for SMPP
Specificity | through the hospitalization, an average of 7 days
  Specificity of prediction model for SMPP
Positive prediction value (PPV) | through the hospitalization, an average of 7 days
  Positive prediction value (PPV) of prediction model for SMPP
Negative prediction value (NPV) | through the hospitalization, an average of 7 days
  Negative prediction value (NPV) of prediction model for SMPP

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided